CLINICAL TRIAL: NCT04795388
Title: Development of an Artificial Intelligence Algorithm to Identify the Main Risks of Ischemia of Mechanical Intestinal Obstruction
Brief Title: Development of an Artificial Intelligence Algorithm
Acronym: SMARTLOOP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SMARTLOOP
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Mechanical Intestinal Obstruction
Keywords: ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical obstruction of the small intestine is an interruption of intestinal transit due to an organic obstacle in the digestive tract that results in a shutdown of materials and gas. Without medical care, it can lead to perforation of the intestinal wall and acute peritonitis. It accounts for 4% of emergency department admissions and 20% of emergency surgeries

DETAILED DESCRIPTION:
The abdominopelvic tomodensitometric examination is the gold standard for making a diagnosis and identifying the cause, the level of the lesion and looking for signs of severity related to the risk of ischemia of the intestinal tissue. Well characterized, these signs remain difficult to identify for a non-expert radiologist. The evaluation of the detection performance of these signs shows a sensitivity between 63 and 100% and a specificity between 61 and 96% with a great variation according to the signs studied.

Our research project aims to develop a tool for the detection of the three main signs of severity of mechanical intestinal obstruction to raise and standardize the level of detection of the risk of ischemia on abdominal CT images.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patients with an abdominal scan performed at Saint-Joseph Hospital
* Patients diagnosed with mechanical obstruction of the small intestine on a flange or adhesion
* Patients having abdominal surgery within 48 hours of diagnosis or medical follow-up at Saint Joseph Hospital
* French-speaking patient

Exclusion Criteria:

* Patients with a history of abdominal surgery one month before diagnosis
* Patients objecting to the use of their data for this research
* Patient under guardianship or curatorship
* Patient under legal protection
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an abdominal scan performed at Saint-Joseph Hospital and diagnosed with mechanical obstruction of the small intestine on a flange or adhesion
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Develop a computer tool that can support the radiologist in identifying the serious risks associated with intestinal obstruction | Day 1
  The comparison score (Dice) between manual classifications and locations performed by clinical experts and those automatically predicted by the tool.
Develop a computer tool that can support the radiologist in identifying the serious risks associated with intestinal obstruction | Day 1
  The number of occlusions

CONTACTS AND LOCATIONS:
Overall Officials: Marc ZINS, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region, France